CLINICAL TRIAL: NCT05134181
Title: Ultrasound Guided Intra-sacroiliac Joint Injection: Methylprednisolone Versus Triamcinolone
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS 20.07.1195
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Sacroiliac Joint Arthritis
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MTP (Active Comparator): will receive ultrasound-guided intra-articular SIJ injection with 40 mg of methylprednisolone with a uniform dose of 2 mL of 2% lidocaine hydrochloride.
  Interventions: Drug: sacroiliac joint injection
- - Group TMC (Active Comparator): will receive ultrasound-guided intra-articular SIJ injection with 40 mg of Triamcinolone acetonide with a uniform dose of 2 mL of 2% lidocaine hydrochloride .
  Interventions: Drug: sacroiliac joint injection

INTERVENTIONS:
Drug: sacroiliac joint injection — Intervention will be done at complete aseptic conditions by ultrasound at frequency of 4-5 MHz patient in prone position. The ultrasound transducer will be oriented in a transverse orientation at the level of the sacral hiatus. Here the sacral cornuae are identified. Moving the transducer laterally from here, the lateral edge of the sacrum is now identified. This bony edge is
  followed in a cephalad direction with the transducer maintained in a transverse orientation. A second bony contour, the ileum, is now identified. The cleft between both bony contours represented the sacroiliac joint. This will be found at 4.5 cm depth. Real-time imaging will be used to direct a 22G spinal needle into the SIJ, where 2% lidocaine and triamcinolone or methylprednisolone will be injected under direct vision.The needle will be removed, a sterile dressing will be applied

SUMMARY:
Intra-articular steroids have been also practiced since a long time. These agents have a better and safer profile as compared to oral drugs in terms of adverse effects/contraindications of the later. Moreover, Intra-articular steroids impart a better pain relief by delivering and also delays any surgical intervention thereby improving the patient's quality of life.

Without imaging, intra-articular injection has been shown in only 22% of patients so ultrasound, fluoroscopic imaging and computerized tomographic (CT) are required to ensure accuracy. Comparing to other guidance, ultrasound guided injection provides easy, safe, accurate, non-invasive, inexpensive imaging and lacking exposure to radiation.

DETAILED DESCRIPTION:
Technique of ultrasound-guided intra-articular SIJ injection:

On arrival to recovery room, an IV line will be secured, ringer solution will be infused, O2 mask with 3l/min oxygen will be supplemented and RBS will be measured. Intervention will be done at complete aseptic conditions by ultrasound at frequency of 4-5 MHz patient in prone position. The ultrasound transducer will be oriented in a transverse orientation at the level of the sacral hiatus. Here the sacral cornuae are identified. Moving the transducer laterally from here, the lateral edge of the sacrum is now identified. This bony edge is

followed in a cephalad direction with the transducer maintained in a transverse orientation. A second bony contour, the ileum, is now identified. The cleft between both bony contours represented the sacroiliac joint. This will be found at 4.5 cm depth. Real-time imaging will be used to direct a 22G spinal needle into the SIJ, where 2% lidocaine and triamcinolone or methylprednisolone will be injected under direct vision.The needle will be removed, a sterile dressing will be applied .then patient lay down at supine position at least 30 minutes with blood pressure ,pulse ,O2 saturation and adverse effect monitoring .

If the pain will be ≥ 4, NSAID will be given to control the pain in the form of 20 mg piroxicam once daily after meal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 - 70 years of both gender,
* sacroiliac pain with at least 3 of the 5 provocative tests are positive,
* pain did not relieved by the conservative therapy (rest, ice/heat, topical menthol, lidocaine patch, pelvic belt, physical therapy and NSIAD) for 4 weeks,
* positive diagnostic test 2 ml lidocaine 2% intra-articular SIJ injection one day before the procedure are included in this study.

Exclusion Criteria:

* The exclusion criteria are patient refusal,
* history of immunosuppression diseases,
* bleeding or coagulation disorders,
* sacroiliac pain of multiple sources,
* local skin infection,
* septic joint, osteomyelitis,
* renal patients (Serum Creatinine >1.8 ),
* decompensated liver diseases,
* local malignancy,
* psychiatric disorders affecting co-operation,
* previous history of chronic opioid use,
* intra articular sacroiliac injection within previous three months,
* negative diagnostic test,
* allergy or hypersensitivity to any of the study medications
* diabetes mellitus, type II with history of poor glycemic control
* morbid obesity ( BMI> 40 ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale at rest and during motion (standing up from a seated position, during stair climbing and walking) | before injection
  numerical rating scale from 0 = no pain to 10 maximum pain
numerical rating scale at rest and during motion (standing up from a seated position, during stair climbing and walking) | after 2 weeks from injection
  numerical rating scale from 0 = no pain to 10 maximum pain
numerical rating scale at rest and during motion (standing up from a seated position, during stair climbing and walking) | after 1 month from injection
  numerical rating scale from 0 = no pain to 10 maximum pain
numerical rating scale at rest and during motion (standing up from a seated position, during stair climbing and walking) | after 2 months from injection
  numerical rating scale from 0 = no pain to 10 maximum pain
numerical rating scale at rest and during motion (standing up from a seated position, during stair climbing and walking) | after 3 months from injection
  numerical rating scale from 0 = no pain to 10 maximum pain

SECONDARY OUTCOMES:
Quality of life | before injection
  Euroqol group 5 dimension 5 level (EQ-5D-5L) questionnaire
Quality of life | after one month of injection
  Euroqol group 5 dimension 5 level (EQ-5D-5L) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Yahya Wahba, Al Mansurah, Egypt